CLINICAL TRIAL: NCT00381056
Title: The Labor and Delivery Teamwork Intervention Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Dynamics Research Corporation (Industry); Armed Forces Institute of Pathology (U.S. Federal Agency); TRICARE Management Activity (Unknown); Harvard Risk Management Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: 2002-P-000044; DAMD171-C-0052
Record Dates: First submitted 2006-09-26; First posted 2006-09-27 (Estimated); Last update posted 2006-09-27 (Estimated); Status verified 2006-09

CONDITIONS: Adverse Maternal and Neonatal Outcomes
Keywords: labor and delivery care; teamwork training; crew resource management; cluster-randomized trial

INTERVENTIONS:
Behavioral: Labor and Delivery Team Coordination Course

SUMMARY:
A cluster-randomized controlled trial was conducted at 7 intervention and 8 control hospitals to evaluate the effect of teamwork training on the occurrence of adverse outcomes and processes of care in labor and delivery.

DETAILED DESCRIPTION:
A cluster-randomized controlled trial was conducted at 7 intervention and 8 control hospitals to evaluate the effect of teamwork training on the occurrence of adverse outcomes and processes of care in labor and delivery. The intervention, called the Labor & Delivery Team Coordination Course, was a standardized teamwork training curriculum based on crew resource management that emphasized communication and team structure. The primary outcome was the proportion of deliveries at greater than or equal to 20 weeks gestation in which one or more adverse maternal and/or neonatal outcomes occurred (Adverse Outcome Index, AOI). Additional outcomes included 11 clinical process measures.

ELIGIBILITY:
Inclusion Criteria:

* delivery at a participating hospital between 12/31/02-03/31/04
* pregnancy of 20-43 weeks gestation

Exclusion Criteria:

* delivery at less than 20 weeks or greater than 43 weeks

Min Age: 0 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30000
Dates: Start 2000-07; Study Completion 2004-03

PRIMARY OUTCOMES:
The primary outcome was the proportion of deliveries at greater than or equal to 20 weeks gestation in which one or more adverse maternal and/or neonatal outcomes occurred (Adverse Outcome Index).

SECONDARY OUTCOMES:
Additional outcomes were eleven process measures that recorded length of care or delay to action.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin P Sachs, MB, BS, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (15):
- United States (15):
  - University of Alabama, Birmingham, Alabama
  - Naval Hospital Campe Pendleton, Oceanside, California
  - Naval Medical Center San Diego, San Diego, California
  - Baptist Health South Florda, Miami, Florida
  - University of Miami, Miami, Florida
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Johns Hopkins Hospital, Baltimore, Maryland
  - National Naval Medical Center Bethesda, Bethesda, Maryland
  - Baystate Hospital, Springfield, Massachusetts
  - South Shore Hospital, Weymouth, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Beaumont Hospital, Royal Oaks, Michigan
  - University of Vermont, Burlington, Vermont
  - Naval Medical Center Portsmouth, Portsmouth, Virginia
  - Madigan Army Medical Center, Tacoma, Washington

REFERENCES:
- [Derived] Nielsen PE, Goldman MB, Mann S, Shapiro DE, Marcus RG, Pratt SD, Greenberg P, McNamee P, Salisbury M, Birnbach DJ, Gluck PA, Pearlman MD, King H, Tornberg DN, Sachs BP. Effects of teamwork training on adverse outcomes and process of care in labor and delivery: a randomized controlled trial. Obstet Gynecol. 2007 Jan;109(1):48-55. doi: 10.1097/01.AOG.0000250900.53126.c2. PMID 17197587